CLINICAL TRIAL: NCT03913338
Title: A Controlled Evaluation of the Safety and Efficacy of Laser In-situ Keratomileusis With Crosslinking (XtraLASIK) Compared to Conventional LASIK (convLASIK) in Patients With High Myopia
Brief Title: Laser In-situ Keratomileusis With Crosslinking Compared to Conventional LASIK in Patients With High Myopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Clinic Frankfurt (Other)
Collaborators: Glaukos Corporation (Industry)
Responsible Party: Principal Investigator, Professor Dr. med. Thomas Kohnen, Head of Ophthalmology, Principal Investigator, Clinical Professor, University Clinic Frankfurt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 154/14
Record Dates: First submitted 2019-04-03; First posted 2019-04-12 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Myopia; Myopic Astigmatism; Crosslinking; Corneal Ectasia; Myopic Regression
MeSH Terms: conditions — Myopia; Astigmatism | interventions — Keratomileusis, Laser In Situ

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, intra-patient controlled, clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Other): LASIK followed by intraoperative application of riboflavin under the flap and crosslinking after reposition of the flap.
  Interventions: Procedure: LasikXtra
- Control group (Other): LASIK only
  Interventions: Procedure: LASIK

INTERVENTIONS:
Procedure: LasikXtra — By randomized selection, one eye was treated with the LASIK Xtra procedure that consists of fs-LASIK treatment combined with intraoperative accelerated continuous UV-riboflavin crosslinking. After laser ablation, the corneal bed under the flap was coated with riboflavin, rinsed with saline solution, and after 90 seconds the corneal flap was repositioned. The eye was irradiated at 30 mW/cm2 for 90 seconds with continuous UVA.
  Arms: Study group
Procedure: LASIK — Femtosecond-assisted preparation of a corneal flap and subsequently excimer-laser ablation of corneal stroma. Repositioning of the corneal flap and installation of a therapeutic contact lens.
  Arms: Control group

SUMMARY:
The objectives of this study are to evaluate the safety and efficacy of a treatment regimen for high myopia and myopic astigmatism: LASIK followed by crosslinking performed with the KXL Crosslinking-System and VibeX Xtra (Riboflavin Ophthalmic Solution, Avedro, USA), as compared to LASIK alone, with regards to regression of refractive outcome, as measured by manifest refraction spherical equivalent (MRSE) and keratometry.

DETAILED DESCRIPTION:
This is a controlled study of the safety and efficacy of the KXL System and VibeX Xtra (Riboflavin Ophthalmic Solution, Avedro, USA) for performing crosslinking in eyes undergoing LASIK for high myopia or myopic astigmatism. Each subject will have bilateral LASIK performed and one eye will be randomized to undergo LASIK followed by crosslinking.

Subjects will undergo bilateral LASIK. Following randomisation one eye of each subject will be treated with VibeX Xtra (Riboflavin Ophthalmic Solution) following LASIK and will be irradiated with the KXL System at 30 mW/cm2 intensity for 90 seconds continuous UV-A light treatment for a total radiant exposure of 2.7 J /cm2.

All eyes will be assessed at 1 day, 1, 3, 6, and 12 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* eligible for bilateral myopic fs-LASIK with -6.00 to -12.00 D (diopters) with a maximum of 5.00 D astigmatism
* age > 18 years
* provided written informed consent
* difference between the MRSE and cycloplegic SE less than 0.75 D
* MRSE needed to be stable for the last 12 months (<0.5 D).

Exclusion Criteria:

* prior corneal surgery,
* forme fruste or manifest keratoconus,
* history of corneal scarring, melting, ulceration
* repeating inflammations of the eye
* taking vitamin C 1 week prior to the treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-07-24 (Actual); Primary Completion 2018-07-03 (Actual); Study Completion 2018-07-03 (Actual)

PRIMARY OUTCOMES:
uncorrected distant visual acuity | 12 months postoperative
  uncorrected distant visual acuity (logarithmic minimum angle of resolution)
best spectacle corrected distant visual acuity | 12 months postoperative
  best spectacle corrected distant visual acuity (logarithmic minimum angle of resolution)
spherical equivalent | 12 months postoperative
  spherical equivalent (diopter)

SECONDARY OUTCOMES:
endothelial cell count | 12 months postoperative
  endothelial cell count (number of cells/ mm2)
Corneal thickness | 12 months postoperative
  Corneal thickness (micro millimeter)
Subjective visual quality | 12 months postoperative
  Questionnaire regarding subjective optical quality (scale from 0 - 100; 0 = minimal, 100 = maximum)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kohnen, Prof. Dr., Principal Investigator — Augenklinik des Universitätsklinikum der Goethe Unveristät Frankfurt am Main
Locations (1):
- Department of ophthalmology University clinic Frankfurt, Frankfurt am Main, Hesse, Germany